CLINICAL TRIAL: NCT01564355
Title: The Role of Postoperative Systemic Corticosteroids When Utilizing a Steroid-Eluting Middle Meatal Spacer Following Endoscopic Sinus Surgery: A Randomized, Double-Blind, Placebo Controlled Trial
Brief Title: Postoperative Systemic Corticosteroids When Utilizing a Steroid-Eluting Spacer Following Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Luke Rudmik, Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24336
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Sinusitis; Endoscopic Sinus Surgery; Post-operative Care; Steroids; Drug-eluting Spacer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Systemic Steroid Group (Experimental): Will receive post-operative oral steroids for 10 days as per usual protocol.
  Interventions: Device: Steroid-eluting middle meatal spacer (Nasopore (TM) spacer impregnated with 1 cc of 40mg/mL triamcinolone liquid); Drug: Post-op Oral Steroids
- Placebo (Placebo Comparator): Will receive placebo pills for 10 days post-operatively
  Interventions: Device: Steroid-eluting middle meatal spacer (Nasopore (TM) spacer impregnated with 1 cc of 40mg/mL triamcinolone liquid)

INTERVENTIONS:
Device: Steroid-eluting middle meatal spacer (Nasopore (TM) spacer impregnated with 1 cc of 40mg/mL triamcinolone liquid) — All study arms will receive bilateral Nasopore spacers impregnated with 1 cc of Triamcinolone to remain in the nasal cavity for 1 week post-operatively as per usual protocol.
Drug: Post-op Oral Steroids — Post-operative oral prednisone 20 mg QD x 5 days , then 10 mg x 5 days, as per usual protocol.
  Arms: Systemic Steroid Group

SUMMARY:
Chronic rhinosinusitis (CRS) is an inflammatory condition of the nose and sinuses. It affects about 5 to 10% of Canadians. Patients suffer from congestion in the nose and sinuses, nasal discharge, pressure in the face, and a reduced sense of smell. This affects people's enjoyment of life. Medical management uses sprays or pills to treat these symptoms but for some patients sinus surgery is needed. This type of surgery is called endoscopic sinus surgery (ESS).

There is no single correct approach to take care of patients after sinus surgery. Most experts would use a nasal spray and a short-course of oral steroid pills to reduce sinus swelling and minimize complications related to scarring.

"Steroid-eluting nasal spacers" are devices placed inside the sinus during surgery and slowly release topical steroids into the sinuses better than steroid sprays. These "spacers" have been shown to improve results following sinus surgery. When using these special "spacers", there may no longer be a need for oral steroid pills following surgery. This would help to avoid potential side effects associated with these medications.

The purpose of this study is to find out whether taking oral (systemic) steroid pills following sinus surgery is necessary to improve surgical results, now that steroid-eluting nasal spacers are commonly used during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult ( > 18 years of age)
* CRS defined by 2007 Adult Sinusitis Guidelines19
* Electing endoscopic sinus surgery for the indication medically refractory CRS, as defined by having persistent symptoms despite the following "maximal medical therapy":

  1. Received 3 months of topical corticosteroid spray
  2. Received a 2 week course of a broad-spectrum antibiotic combined with a 2 week course of systemic corticosteroid
* Provide written informed consent
* Subject must be able to complete all study evaluations and HRQoL questionnaires written in English

Exclusion Criteria:

* Children (< 18 years of age)
* Unable to complete questionnaires or clinical testing or cooperate with study evaluations in English.
* Unwilling to provide written, informed consent
* Patients who have not undergone previous "maximum" prescribed medical therapy
* Patients with suspected systemic inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life Score (based on SNOT-22, VAS, and RSDI questionnaires) | Up to 2 years
  Do systemic steroids following sinus surgery improve surgical results in patients where a steroid-eluting nasal spacer is placed at the completion of surgery. This will be based on validated chronic sinusitis-symptom specific HRQOL questionnaires (SNOT-22, VAS, RSDI)and mucosal disease grading scores via endoscopic examination (POSE, Lund-Kennedy).

SECONDARY OUTCOMES:
Sinus mucosal disease endoscopic grading score (based on Lund-Kennedy and POSE Scoring systems) | Up to 3 years
  Do systemic steroids following sinus surgery improve surgical results in patients where a steroid-eluting nasal spacer is placed at the completion of surgery. This will be based on validated mucosal disease grading scores via endoscopic examination (POSE, Lund-Kennedy).

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Road Diagnostic and Treatment Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Dautremont JF, Mechor B, Rudmik L. The role of immediate postoperative systemic corticosteroids when utilizing a steroid-eluting spacer following sinus surgery. Otolaryngol Head Neck Surg. 2014 Apr;150(4):689-95. doi: 10.1177/0194599814521373. Epub 2014 Jan 30. PMID 24482348